CLINICAL TRIAL: NCT01128569
Title: A Randomised, Double-blind, Placebo-controlled, Three-way Crossover, Repeat Dose Pilot Study Comparing the Effect of Inhaled Fluticasone Furoate/GW642444M Combination and Fluticasone Furoate on the Allergen-induced Early Asthmatic Response in Subjects With Mild Asthma
Brief Title: Randomised Study Comparing the Effects of Inhaled Fluticasone Furoate (FF)/Vilanterol (VI; GW642444M) Combination and FF on an Allergen Induced Asthmatic Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 113090
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Results first posted 2013-09-11 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: mild asthma; allergen challenge; early asthmatic response
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo Inhaler
  Interventions: Drug: Placebo
- inhaled corticosteroid(ICS)/long acting bronchodilator (LABA) (Active Comparator): ICS/LABA inhaler
  Interventions: Drug: FF/Vilanterol (VI; GW642444M)
- ICS (Active Comparator): ICS inhaler
  Interventions: Drug: Fluticasone Furoate

INTERVENTIONS:
Drug: Fluticasone Furoate — FF
  Other Names: FF
  Arms: ICS
Drug: FF/Vilanterol (VI; GW642444M) — FF/VI
  Other Names: FF/VI
  Arms: inhaled corticosteroid(ICS)/long acting bronchodilator (LABA)
Drug: Placebo — Placebo Inhaler
  Arms: Placebo

SUMMARY:
We propose to use an inhaled allergen challenge model to explore the individual contributions of the components of a novel long-acting beta agonist (LABA)/ inhaled corticosteroid (ICS) combination product on protection from allergic triggers in asthma.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index within the range 18.5-35.0 kilograms/metre2 (kg/m2).
* Females of non-child bearing potential.
* Documented history of bronchial asthma, first diagnosed at least 6 months prior to the screening visit and currently being treated only with intermittent short-acting beta -agonist therapy by inhalation
* Pre-bronchodilator FEV1 >70% of predicted at screening
* Subjects who are current non-smokers
* Methacholine challenge PC20 < 8 mg/mL at screening
* Screening allergen challenge demonstrates that the subject experiences an early asthmatic response

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* Subject is hypertensive at screening
* Respiratory tract infection and/or exacerbation of asthma within 4 weeks prior to the first dose of study medication.
* History of life-threatening asthma
* Symptomatic with hay fever at screening or predicted to have symptomatic hayfever
* Unable to abstain from short acting beta agonists
* Unable to abstain from antihistamines
* Unable to abstain from other medications including non-steroidal anti-inflammatory drugs (NSAIDs), anti-depressant drugs, anti-asthma anti-rhinitis or hay fever medication
* The subject has participated in a study with a new molecular entity during the previous 3 months or has participated in 4 or more clinical studies in the previous 12 months
* undergoing allergen desensitisation therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Berlin, State of Berlin, Germany
- GSK Investigational Site, Wellington, New Zealand
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Oliver A, Quinn D, Goldfrad C, van Hecke B, Ayer J, Boyce M. Combined fluticasone furoate/vilanterol reduces decline in lung function following inhaled allergen 23 h after dosing in adult asthma: a randomised, controlled trial. Clin Transl Allergy. 2012 Jun 27;2(1):11. doi: 10.1186/2045-7022-2-11. PMID 22738148
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 113090 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113090 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113090 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113090 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113090 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113090 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113090 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened within 42 days of the first dose, conducted over 2 days (not consecutive days). During this time, a methacholine challenge and an allergen challenge test were performed. Participants meeting all inclusion criteria and none of the exclusion criteria were randomized to 3 study treatment periods, each lasting 28 days.
Pre-assignment Details: This study was a multi-center, randomized, double-blind, placebo controlled, three-period crossover study in mild asthmatic male and female participants. Following the Run-in period, participants were randomized to 1 of 6 treatment sequences of placebo, FF 100 micrograms (µg) once daily (OD), and FF/VI 100/25 µg OD.
Groups:
- Sequence 1: Placebo, FF 100 µg, FF/VI 100/25 µg: Participants received placebo, Fluticasone Furoate (FF) 100 micrograms (µg), and FF/Vilanterol (VI) 100/25 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments once a day (OD) in the evening from a Dry Powder Inhaler (DPI) for 28 days. The three treatment periods were separated by a washout period of at least 21 days (from the Day 28 dose) and a maximum of 35 days.
- Sequence 2: Placebo, FF/VI 100/25 µg, FF 100 µg: Participants received placebo, FF/VI 100/25 µg, and FF 100 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments once a day in the evening from a DPI for 28 days. The three treatment periods were separated by a washout period of at least 21 days (from the Day 28 dose) and a maximum of 35 days.
- Sequence 3: FF 100 µg, FF/VI 100/25 µg, Placebo: Participants received FF 100 µg, FF/VI 100/25 µg, and placebo in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments once a day in the evening from a DPI for 28 days. The three treatment periods were separated by a washout period of at least 21 days (from the Day 28 dose) and a maximum of 35 days.
- Sequence 4: FF 100 µg, Placebo, FF/VI 100/25 µg: Participants received FF 100 µg, placebo, and FF/VI 100/25 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments once a day in the evening from a DPI for 28 days. The three treatment periods were separated by a washout period of at least 21 days (from the Day 28 dose) and a maximum of 35 days.
- Sequence 5: FF/VI 100/25 µg, Placebo, FF 100 µg: Participants received FF/VI 100/25 µg, placebo, and FF 100 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments once a day in the evening from a DPI for 28 days. The three treatment periods were separated by a washout period of at least 21 days (from the Day 28 dose) and a maximum of 35 days.
- Sequence 6: FF/VI 100/25 µg, FF 100 µg, Placebo: Participants received FF/VI 100/25 µg, FF 100 µg, and placebo in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments once a day in the evening from a DPI for 28 days. The three treatment periods were separated by a washout period of at least 21 days (from the Day 28 dose) and a maximum of 35 days.
Period: Treatment Period 1
Arm/Group | Sequence 1: Placebo, FF 100 µg, FF/VI 100/25 µg | Sequence 2: Placebo, FF/VI 100/25 µg, FF 100 µg | Sequence 3: FF 100 µg, FF/VI 100/25 µg, Placebo | Sequence 4: FF 100 µg, Placebo, FF/VI 100/25 µg | Sequence 5: FF/VI 100/25 µg, Placebo, FF 100 µg | Sequence 6: FF/VI 100/25 µg, FF 100 µg, Placebo
Started | 9 | 8 | 9 | 8 | 9 | 9
Completed | 9 | 8 | 9 | 8 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Sequence 1: Placebo, FF 100 µg, FF/VI 100/25 µg | Sequence 2: Placebo, FF/VI 100/25 µg, FF 100 µg | Sequence 3: FF 100 µg, FF/VI 100/25 µg, Placebo | Sequence 4: FF 100 µg, Placebo, FF/VI 100/25 µg | Sequence 5: FF/VI 100/25 µg, Placebo, FF 100 µg | Sequence 6: FF/VI 100/25 µg, FF 100 µg, Placebo
Started | 9 | 8 | 9 | 8 | 9 | 9
Completed | 9 | 8 | 8 | 8 | 9 | 9
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Sequence 1: Placebo, FF 100 µg, FF/VI 100/25 µg | Sequence 2: Placebo, FF/VI 100/25 µg, FF 100 µg | Sequence 3: FF 100 µg, FF/VI 100/25 µg, Placebo | Sequence 4: FF 100 µg, Placebo, FF/VI 100/25 µg | Sequence 5: FF/VI 100/25 µg, Placebo, FF 100 µg | Sequence 6: FF/VI 100/25 µg, FF 100 µg, Placebo
Started | 9 | 8 | 8 | 8 | 9 | 9
Completed | 9 | 7 | 8 | 8 | 9 | 9
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Sequence 1: Placebo, FF 100 µg, FF/VI 100/25 µg | Sequence 2: Placebo, FF/VI 100/25 µg, FF 100 µg | Sequence 3: FF 100 µg, FF/VI 100/25 µg, Placebo | Sequence 4: FF 100 µg, Placebo, FF/VI 100/25 µg | Sequence 5: FF/VI 100/25 µg, Placebo, FF 100 µg | Sequence 6: FF/VI 100/25 µg, FF 100 µg, Placebo
Started | 9 | 7 | 8 | 8 | 9 | 9
Completed | 9 | 7 | 8 | 8 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Sequence 1: Placebo, FF 100 µg, FF/VI 100/25 µg | Sequence 2: Placebo, FF/VI 100/25 µg, FF 100 µg | Sequence 3: FF 100 µg, FF/VI 100/25 µg, Placebo | Sequence 4: FF 100 µg, Placebo, FF/VI 100/25 µg | Sequence 5: FF/VI 100/25 µg, Placebo, FF 100 µg | Sequence 6: FF/VI 100/25 µg, FF 100 µg, Placebo
Started | 9 | 7 | 8 | 8 | 9 | 9
Completed | 9 | 7 | 8 | 8 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo, FF 100 µg OD, FF/VI 100/25 µg OD in 1 of 6 Sequences: All participants received one of the following three treatments in one of three treatment periods once daily (OD) in the evening from the Dry Powder Inhaler (DPI) for 28 days: Placebo, Fluticasone Furoate (FF) 100 microgram (µg) dry inhalation powder, and FF/Vilanterol (FF/VI) 100/25 µg dry inhalation powder. Participants were randomized to receive treatment in one of the six following sequences: (1) Placebo, FF 100 µg, FF/VI 100/25 µg; (2) Placebo, FF/VI 100/25 µg, FF 100 µg; (3) FF 100 µg, FF/VI 100/25 µg, Placebo; (4) FF 100 µg, Placebo, FF/VI 100/25 µg; (5) FF/VI 100/25 µg, Placebo, FF 100 µg; (6) FF/VI 100/25 µg, FF 100 µg, Placebo. The three treatment periods were separated by a washout period of at least 21 days (from the Day 28 dose) and a maximum of 35 days.
Arm/Group | Placebo, FF 100 µg OD, FF/VI 100/25 µg OD in 1 of 6 Sequences
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.4 (8.63)
Gender [Count of Participants; unit: Participants]
  Female | 18
  Male | 34
Race/Ethnicity, Customized [Number; unit: participants]
  White - White/Caucasian/European Heritage | 48
  African American/African Heritage | 2
  Asian - South East Asian Heritage | 1
  Mixed Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Weighted Mean Change From Baseline in Forced Expiratory Volume in One Second (FEV1) Between 0-2 Hours, Following the 22-23 Hour Post-treatment Allergen Challenge on Day 29 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants (par.) were exposed to an allergen (administered by inhalation) 22-23 hours after dosing on Day 28. FEV1 was measured 5 minutes (min), 10 min, 15 min, 20 min, 30 min, and 45 min and 1 hour, 1.5 hours, and 2 hours post-allergen challenge on Day 29. Immediately prior to the exposure of allergen and starting at 2 minutes after inhalation of saline, 3 single measurements of FEV1 were recorded at 1-minute intervals, and the best was taken as the post-saline value. The FEV1 weighted mean was derived by calculating the area under the curve, and then dividing the value by the relevant time interval. Weighted mean change from Baseline is calculated as the weighted mean FEV1 value on Day 29 minus the Baseline value. The Baseline FEV1 value was the post-saline value on Day 29.
Time Frame: Baseline and Day 29 of each treatment period (up to Study Day 197)
Population: Intent-to-Treat (ITT) Population: par. randomized to treatment who received >=1 dose of study drug. Only those par. available at the specified time points were analyzed. Analysis was performed using mixed model analysis of covariance (ANCOVA) with fixed effects of treatment, period, par.-level Baseline, period level Baseline, country, sex, and age.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Placebo: Participants received Placebo OD from the DPI in the evening for 28 days during one of the three treatment periods. Each treatment period was followed by a washout of at least 21 days (from the Day 28 dose) and a maximum of 35 days.
- FF 100 µg OD: Participants received FF 100 µg dry inhalation powder OD in the evening from the DPI for 28 days during one of the three treatment periods. Each treatment period was followed by a washout of at least 21 days (from Day 28 dose) and a maximum of 35 days.
- FF/VI 100/25 µg OD: Participants received FF/VI 100/25 µg dry inhalation powder OD from the DPI in the evening for 28 days during one of the three treatment periods. Each treatment period was followed by a washout of at least 21 days (from Day 28 dose) and a maximum of 35 days.
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 45 | 49 | 46
Liters | -0.372 (0.0557) | -0.210 (0.0549) | -0.227 (0.0550)
Statistical Analysis 1: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.162, 95% CI 2-sided [0.087 to 0.237]
Statistical Analysis 2: Comparison: Placebo vs FF/VI 100/25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.145, 95% CI 2-sided [0.069 to 0.222]
Statistical Analysis 3: Comparison: FF 100 µg OD vs FF/VI 100/25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.017, 95% CI 2-sided [-0.091 to 0.057]

2. Secondary Outcome: Maximum Percent Decrease From Baseline in FEV1 Between 0 2 Hour, Following the 22-23 Hour Post-treatment Allergen Challenge on Day 29 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants were exposed to an allergen 22-23 hours after dosing on Day 28. Immediately prior to the exposure of allergen and starting at 2 minutes (min) after inhalation of saline, 3 single measurements of FEV1were recorded at 1-min intervals, and the best was taken as the post-saline value. The maximum change (i.e., drop in FEV1) from post-saline Baseline (BL) is defined by ordering all of the change from BL values for the 5 min, 10 min, 15 min, 20 min, 30 min, and 45 min and the 1 hour, 1.5 hours, and 2 hours post-allergen challenge and selecting the largest change (i.e., drop in FEV1) from the BL value. If there were no negative change values, indicating a worse FEV1 value as compared to the BL value, the smallest change in FEV1, indicating an improvement from the BL value, was selected. The BL FEV1 value was the post-saline value on Day 29.
Time Frame: Baseline and Day 29 of each treatment period (up to Study Day 197)
Population: ITT Population. Only those participants available at the specified time points were analyzed. Analysis was performed using mixed model analysis of covariance (ANCOVA) with fixed effects of treatment, period, participant-level BL, period level BL, country, sex, and age. Change from BL was calculated as the value on Day 29 minus the BL value.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 45 | 49 | 46
Percent change | -24.991 (2.0736) | -14.040 (2.0435) | -13.206 (2.0491)

3. Secondary Outcome: Minimum FEV1 Absolute Change From Baseline Between 0-2 Hour, Following the 22-23 Hour Post-treatment Allergen Challenge on Day 29 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants were exposed to an allergen 22-23 hours after dosing on Day 28. Immediately prior to the exposure of allergen and starting at 2 minutes after inhalation of saline, 3 single measurements of FEV1were recorded at 1-minute intervals, and the best was taken as the post-saline value. The minimum FEV1 over 0-2 hours post-allergen challenge (PAC) (minimum early asthmatic response) was the minimum value of all of the PAC time points up to and including 2 hours PAC (i.e., minimum over 5 minutes (min), 10 min, 15 min, 20 min, 30 min, and 45 min and 1 hour, 1.5 hours, and 2 hours). Change from Baseline was calculated using the post-saline FEV1 on Day 29 as Baseline. Minimum FEV1 absolute change from Baseline between 0-2 hour, following the 22-23 hour post-treatment allergen challenge was calculated as the minimum change value on Day 29 minus the Baseline value
Time Frame: Baseline and Day 29 of each treatment period (up to Study Day 197)
Population: ITT Population. Only those participants available at the specified time points were analyzed. Analysis was performed using mixed model ANCOVA with fixed effects of treatment, period, participant-level Baseline, period level Baseline, country, sex, and age.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 45 | 49 | 46
Liters | -0.809 (0.0775) | -0.479 (0.0765) | -0.478 (0.0767)

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs)
Description: The number of participants with treatment-emergent AEs was measured. A treatment-emergent adverse event is defined as any event not present prior to the initiation of the treatments, or any event already present that worsens in either intensity of frequency following exposure to the treatments.
Time Frame: From the start of study medication until Follow-up/Early Withdrawal (up to 197 days)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Number analyzed (Participants) | 51 | 51 | 51
participants | 20 | 22 | 18

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication until Follow-up/Early Withdrawal (up to 197 days).
Description: SAEs and non-serious AEs were reported for members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of study drug.
Arm/Group | Placebo | FF 100 µg OD | FF/VI 100/25 µg OD
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 15/51 | 18/51 | 11/51
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | FF 100 µg OD (N=51) | FF/VI 100/25 µg OD (N=51)
Headache (Nervous system disorders) | 9 | 11 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 2 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 0
Chest discomfort (General disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.